CLINICAL TRIAL: NCT03829176
Title: Investigating the Feasibility and Implementation of Whole Genome Sequencing in Patients With Suspected Genetic Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Broad Institute of MIT and Harvard (Other); Laboratory for Molecular Medicine (Unknown)
Responsible Party: Principal Investigator, Sekar Kathiresan, Director of the Center for Genomic Medicine, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 2017P001832
Record Dates: First submitted 2018-10-30; First posted 2019-02-04 (Actual); Last update posted 2020-11-18 (Actual); Status verified 2020-11

CONDITIONS: Hereditary Disease; Genetic Predisposition to Disease
Keywords: Whole Genome Sequencing
MeSH Terms: conditions — Genetic Diseases, Inborn; Genetic Predisposition to Disease | interventions — Whole Genome Sequencing

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: Participant, care provider, and study genetic counselor will be blinded to the arm in which the participant was assigned until 3-4 months post-enrollment when the laboratory notifies if a WGS report is generated or not.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard-of-Care (No Intervention): Participants who are randomized to not have whole genome sequencing performed on their sample. These participants will have standard-of-care genetic testing only (ordered by their clinical provider) and will not receive genetic results as part of this study.
- Whole Genome Sequencing (Experimental): Participants who are randomized to have their genome sequenced and receive a whole genome sequencing report. Results disclosure sessions will include a discussion of the whole genome sequencing report, how the results compare to their standard-of-care genetic testing report, and any potential relevant recommendations. Participants in this arm will receive a copy of their whole genome sequencing report accompanied by a summary letter written by a study genetic counselor.
  Interventions: Genetic: Whole Genome Sequencing

INTERVENTIONS:
Genetic: Whole Genome Sequencing — Participants in this arm will have their sample analyzed by whole genome sequencing (WGS), and a report will be included in their medical record. Analysis will be phenotype-driven (gene list will be curated based on primary indication for testing and other available medical history information), and may include genes on ACMG 59 list if participant elects for these results. This report will include pathogenic, likely pathogenic, and suspicious VUS results identified in the genes analyzed.
  Arms: Whole Genome Sequencing

SUMMARY:
The study "Investigating the Feasibility and Implementation of Whole Genome Sequencing in Patients With Suspected Genetic Disorder" is a research study that aims to explore the use of whole genome sequencing as a potential first line genetic test for patients for which a genetic diagnosis is suspected. This is an internally funded research study.

The investigators will enroll 500 participants who are being seen in one of the various genetics clinics within the Partners HealthCare system for a suspected genetic disorder for which standard-of-care genetic testing is ordered. At the time of their standard-of-care genetic testing, an extra blood sample will be collected, and genome sequencing may be performed. Within 3-4 months, patients learn if they received genome sequencing or not, and any results are returned and explained. Investigators are also studying the experiences of both participants and their providers to better understand how to implement genome sequencing into clinical care.

DETAILED DESCRIPTION:
The goal of this research protocol is to conduct a randomized clinical trial to assess the benefits and risks of incorporating whole genome sequencing (WGS) as a first line diagnostic test in various genetic and sub-specialty clinics within a large, tertiary medical center.

The investigators will enroll 500 participants within the Partners HealthCare system (e.g. Massachusetts General Hospital, Massachusetts Eye and Ear, etc.). The study will be enrolling from multiple genetics and sub-specialty clinics, including but not limited to: cardiology, GI cancer genetics, medical genetics, ataxia, endocrine genetics. Participants are eligible if their provider orders genetic testing for diagnosis of symptoms suspicious for a genetic disorder. Participants must not have had a genetic workup in the past.

At the time of enrollment, a small blood sample will be obtained at the time of the participant's blood draw for standard-of-care testing. All participants will be subject to 1:1 randomization, in which 250 will receive a WGS report, and 250 will be randomized to the arm that receives standard of care testing only. Any WGS report that is generated will be incorporated into the patient's electronic medical record.

For pediatric patients, the study team will attempt to collect blood samples from both biological parents when possible for trio analysis (WGS performed on the proband and both biological parents). The purpose of trio analysis is primarily for the purpose of interpreting the proband/child's results. For non-pediatric patients, saliva samples may be requested from living parents for confirmation purposes. No genetic testing reports will be generated for parents. The exception to this is if a parent of a pediatric patient (part of trio) opts to receive results from the ACMG 59 list.

The participants are blinded to the arm in which they are assigned until 3-4 months from the time of consent. At that time, a study genetic counselor will call the participant to disclose the randomization assignment. If the participant was randomized to receive a WGS report, a plan will be made to review the WGS either by phone, video conferencing, or in person. After reviewing the results, the research team will write a letter to the participant summarizing the results and any relevant medical management recommendations. This letter will also include a copy of their WGS report.

All participants (or their parents) will be surveyed at three points during their enrollment: baseline (at time of consent), immediately post-disclosure, and 6 months post-disclosure. The medical providers who offered the standard of care testing will also be surveyed.

ELIGIBILITY:
Inclusion Criteria:

1. Participants of any gender over the age of 3 months.
2. Participants (ages 7+) must be proficient in English. If the participant is under the age of 7 or is over the age of 7 and non-verbal, these criteria apply to their parent who is providing consent.
3. Participant is being evaluated clinically at an Partners HealthCare genetics clinic, and not had a prior genetic work up for their referral indication.
4. Have a suspected genetic disorder in which the genetic cause is unknown, as confirmed by review of the subject's medical records.
5. Genetic testing has been ordered for the participant by their clinical genetics provider as part of a diagnostic workup.
6. Willing and able to provide a blood sample. The amount of blood drawn from a patient will be 2 teaspoons or less.
7. Ability to provide informed consent or assent to participate in this protocol. Children who have not attained the legal age of consent must provide assent (those who do not have the capacity to assent must not object to taking part), along with permission from the child's parent(s) or guardian. Adults who are unable to consent must be able to provide assent or must not object to taking part, along with permission from their legal authorized representative (LAR).

Exclusion Criteria:

1. Participants who live outside of the United States.
2. Non-English-speaking participants.

Min Age: 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
Diagnostic capabilities: standard-of-care vs whole genome sequencing diagnostic yield | From date of consent until the date of first documented report, assessed up to 12 months
  Assess and compare the overall yields for primary and secondary/incidental findings
Diagnostic capabilities: standard-of-care vs whole genome sequencing time to reach diagnosis | From date of consent until the date of first positive report, assessed up to 12 months
  Assess and compare the time that is required to reach a diagnosis by both standard-of-care genetic testing and whole genome sequencing

SECONDARY OUTCOMES:
Resources Needed to Implement WGS at an Academic Medical Center | Baseline to End of Study, up to 2 years
  Assess by recording resources needed to implement WGS at an Academic Medical Center by documenting resources needed for engagement, execution, reporting, and evaluation.
Participant characteristics | Baseline
  Age, sociodemographics, personal and family history
Change in perceived utility of genomic results | Baseline, post-disclosure (approximately 3-4 months after enrollment), 6 months post-disclosure
  Assessed in participant (or parent) surveys via questions assessing: reasons for decline, motivations for enrollment, change in expectations, confidence, concerns, preferences for information sharing
Physician confidence and attitudes about genomic sequencing | Baseline
  Assessed in physician surveys

CONTACTS AND LOCATIONS:
Overall Officials: Sekar Kathiresan, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Sherman S, Pletcher BA, Driscoll DA. Fragile X syndrome: diagnostic and carrier testing. Genet Med. 2005 Oct;7(8):584-7. doi: 10.1097/01.gim.0000182468.22666.dd. PMID 16247297
- [Background] Ross LF, Saal HM, David KL, Anderson RR; American Academy of Pediatrics; American College of Medical Genetics and Genomics. Technical report: Ethical and policy issues in genetic testing and screening of children. Genet Med. 2013 Mar;15(3):234-45. doi: 10.1038/gim.2012.176. Epub 2013 Feb 21. PMID 23429433
- [Background] Manning M, Hudgins L; Professional Practice and Guidelines Committee. Array-based technology and recommendations for utilization in medical genetics practice for detection of chromosomal abnormalities. Genet Med. 2010 Nov;12(11):742-5. doi: 10.1097/GIM.0b013e3181f8baad. PMID 20962661
- [Background] Xue Y, Ankala A, Wilcox WR, Hegde MR. Solving the molecular diagnostic testing conundrum for Mendelian disorders in the era of next-generation sequencing: single-gene, gene panel, or exome/genome sequencing. Genet Med. 2015 Jun;17(6):444-51. doi: 10.1038/gim.2014.122. Epub 2014 Sep 18. PMID 25232854
- [Background] Yang Y, Muzny DM, Reid JG, Bainbridge MN, Willis A, Ward PA, Braxton A, Beuten J, Xia F, Niu Z, Hardison M, Person R, Bekheirnia MR, Leduc MS, Kirby A, Pham P, Scull J, Wang M, Ding Y, Plon SE, Lupski JR, Beaudet AL, Gibbs RA, Eng CM. Clinical whole-exome sequencing for the diagnosis of mendelian disorders. N Engl J Med. 2013 Oct 17;369(16):1502-11. doi: 10.1056/NEJMoa1306555. Epub 2013 Oct 2. PMID 24088041
- [Background] Lee H, Deignan JL, Dorrani N, Strom SP, Kantarci S, Quintero-Rivera F, Das K, Toy T, Harry B, Yourshaw M, Fox M, Fogel BL, Martinez-Agosto JA, Wong DA, Chang VY, Shieh PB, Palmer CG, Dipple KM, Grody WW, Vilain E, Nelson SF. Clinical exome sequencing for genetic identification of rare Mendelian disorders. JAMA. 2014 Nov 12;312(18):1880-7. doi: 10.1001/jama.2014.14604. PMID 25326637
- [Background] Vissers LELM, van Nimwegen KJM, Schieving JH, Kamsteeg EJ, Kleefstra T, Yntema HG, Pfundt R, van der Wilt GJ, Krabbenborg L, Brunner HG, van der Burg S, Grutters J, Veltman JA, Willemsen MAAP. A clinical utility study of exome sequencing versus conventional genetic testing in pediatric neurology. Genet Med. 2017 Sep;19(9):1055-1063. doi: 10.1038/gim.2017.1. Epub 2017 Mar 23. PMID 28333917
- [Background] de Ligt J, Willemsen MH, van Bon BW, Kleefstra T, Yntema HG, Kroes T, Vulto-van Silfhout AT, Koolen DA, de Vries P, Gilissen C, del Rosario M, Hoischen A, Scheffer H, de Vries BB, Brunner HG, Veltman JA, Vissers LE. Diagnostic exome sequencing in persons with severe intellectual disability. N Engl J Med. 2012 Nov 15;367(20):1921-9. doi: 10.1056/NEJMoa1206524. Epub 2012 Oct 3. PMID 23033978
- [Background] Yang Y, Muzny DM, Xia F, Niu Z, Person R, Ding Y, Ward P, Braxton A, Wang M, Buhay C, Veeraraghavan N, Hawes A, Chiang T, Leduc M, Beuten J, Zhang J, He W, Scull J, Willis A, Landsverk M, Craigen WJ, Bekheirnia MR, Stray-Pedersen A, Liu P, Wen S, Alcaraz W, Cui H, Walkiewicz M, Reid J, Bainbridge M, Patel A, Boerwinkle E, Beaudet AL, Lupski JR, Plon SE, Gibbs RA, Eng CM. Molecular findings among patients referred for clinical whole-exome sequencing. JAMA. 2014 Nov 12;312(18):1870-9. doi: 10.1001/jama.2014.14601. PMID 25326635
- [Background] Gonorazky H, Liang M, Cummings B, Lek M, Micallef J, Hawkins C, Basran R, Cohn R, Wilson MD, MacArthur D, Marshall CR, Ray PN, Dowling JJ. RNAseq analysis for the diagnosis of muscular dystrophy. Ann Clin Transl Neurol. 2015 Dec 8;3(1):55-60. doi: 10.1002/acn3.267. eCollection 2016 Jan. PMID 26783550
- [Background] Meienberg J, Bruggmann R, Oexle K, Matyas G. Clinical sequencing: is WGS the better WES? Hum Genet. 2016 Mar;135(3):359-62. doi: 10.1007/s00439-015-1631-9. Epub 2016 Jan 7. PMID 26742503
- [Background] Taylor JC, Martin HC, Lise S, Broxholme J, Cazier JB, Rimmer A, Kanapin A, Lunter G, Fiddy S, Allan C, Aricescu AR, Attar M, Babbs C, Becq J, Beeson D, Bento C, Bignell P, Blair E, Buckle VJ, Bull K, Cais O, Cario H, Chapel H, Copley RR, Cornall R, Craft J, Dahan K, Davenport EE, Dendrou C, Devuyst O, Fenwick AL, Flint J, Fugger L, Gilbert RD, Goriely A, Green A, Greger IH, Grocock R, Gruszczyk AV, Hastings R, Hatton E, Higgs D, Hill A, Holmes C, Howard M, Hughes L, Humburg P, Johnson D, Karpe F, Kingsbury Z, Kini U, Knight JC, Krohn J, Lamble S, Langman C, Lonie L, Luck J, McCarthy D, McGowan SJ, McMullin MF, Miller KA, Murray L, Nemeth AH, Nesbit MA, Nutt D, Ormondroyd E, Oturai AB, Pagnamenta A, Patel SY, Percy M, Petousi N, Piazza P, Piret SE, Polanco-Echeverry G, Popitsch N, Powrie F, Pugh C, Quek L, Robbins PA, Robson K, Russo A, Sahgal N, van Schouwenburg PA, Schuh A, Silverman E, Simmons A, Sorensen PS, Sweeney E, Taylor J, Thakker RV, Tomlinson I, Trebes A, Twigg SR, Uhlig HH, Vyas P, Vyse T, Wall SA, Watkins H, Whyte MP, Witty L, Wright B, Yau C, Buck D, Humphray S, Ratcliffe PJ, Bell JI, Wilkie AO, Bentley D, Donnelly P, McVean G. Factors influencing success of clinical genome sequencing across a broad spectrum of disorders. Nat Genet. 2015 Jul;47(7):717-726. doi: 10.1038/ng.3304. Epub 2015 May 18. PMID 25985138
- [Background] Gilissen C, Hehir-Kwa JY, Thung DT, van de Vorst M, van Bon BW, Willemsen MH, Kwint M, Janssen IM, Hoischen A, Schenck A, Leach R, Klein R, Tearle R, Bo T, Pfundt R, Yntema HG, de Vries BB, Kleefstra T, Brunner HG, Vissers LE, Veltman JA. Genome sequencing identifies major causes of severe intellectual disability. Nature. 2014 Jul 17;511(7509):344-7. doi: 10.1038/nature13394. Epub 2014 Jun 4. PMID 24896178
- [Background] Stavropoulos DJ, Merico D, Jobling R, Bowdin S, Monfared N, Thiruvahindrapuram B, Nalpathamkalam T, Pellecchia G, Yuen RKC, Szego MJ, Hayeems RZ, Shaul RZ, Brudno M, Girdea M, Frey B, Alipanahi B, Ahmed S, Babul-Hirji R, Porras RB, Carter MT, Chad L, Chaudhry A, Chitayat D, Doust SJ, Cytrynbaum C, Dupuis L, Ejaz R, Fishman L, Guerin A, Hashemi B, Helal M, Hewson S, Inbar-Feigenberg M, Kannu P, Karp N, Kim R, Kronick J, Liston E, MacDonald H, Mercimek-Mahmutoglu S, Mendoza-Londono R, Nasr E, Nimmo G, Parkinson N, Quercia N, Raiman J, Roifman M, Schulze A, Shugar A, Shuman C, Sinajon P, Siriwardena K, Weksberg R, Yoon G, Carew C, Erickson R, Leach RA, Klein R, Ray PN, Meyn MS, Scherer SW, Cohn RD, Marshall CR. Whole Genome Sequencing Expands Diagnostic Utility and Improves Clinical Management in Pediatric Medicine. NPJ Genom Med. 2016 Jan 13;1:15012-. doi: 10.1038/npjgenmed.2015.12. PMID 28567303
- [Background] Vassy JL, Christensen KD, Schonman EF, Blout CL, Robinson JO, Krier JB, Diamond PM, Lebo M, Machini K, Azzariti DR, Dukhovny D, Bates DW, MacRae CA, Murray MF, Rehm HL, McGuire AL, Green RC; MedSeq Project. The Impact of Whole-Genome Sequencing on the Primary Care and Outcomes of Healthy Adult Patients: A Pilot Randomized Trial. Ann Intern Med. 2017 Jun 27;167(3):159-169. doi: 10.7326/M17-0188. Print 2017 Aug 1. PMID 28654958
- [Background] RARE Diseases: Facts and Statistics. (2017, March 29). Retrieved July 19, 2017, from https://globalgenes.org/rare-diseases-facts-statistics/
- [Background] Fullerton SM, Wolf WA, Brothers KB, Clayton EW, Crawford DC, Denny JC, Greenland P, Koenig BA, Leppig KA, Lindor NM, McCarty CA, McGuire AL, McPeek Hinz ER, Mirel DB, Ramos EM, Ritchie MD, Smith ME, Waudby CJ, Burke W, Jarvik GP. Return of individual research results from genome-wide association studies: experience of the Electronic Medical Records and Genomics (eMERGE) Network. Genet Med. 2012 Apr;14(4):424-31. doi: 10.1038/gim.2012.15. Epub 2012 Feb 23. PMID 22361898
- [Background] Kalia SS, Adelman K, Bale SJ, Chung WK, Eng C, Evans JP, Herman GE, Hufnagel SB, Klein TE, Korf BR, McKelvey KD, Ormond KE, Richards CS, Vlangos CN, Watson M, Martin CL, Miller DT. Recommendations for reporting of secondary findings in clinical exome and genome sequencing, 2016 update (ACMG SF v2.0): a policy statement of the American College of Medical Genetics and Genomics. Genet Med. 2017 Feb;19(2):249-255. doi: 10.1038/gim.2016.190. Epub 2016 Nov 17. PMID 27854360
- [Background] Green RC, Berg JS, Grody WW, Kalia SS, Korf BR, Martin CL, McGuire AL, Nussbaum RL, O'Daniel JM, Ormond KE, Rehm HL, Watson MS, Williams MS, Biesecker LG; American College of Medical Genetics and Genomics. ACMG recommendations for reporting of incidental findings in clinical exome and genome sequencing. Genet Med. 2013 Jul;15(7):565-74. doi: 10.1038/gim.2013.73. Epub 2013 Jun 20. PMID 23788249
- [Background] Richards S, Aziz N, Bale S, Bick D, Das S, Gastier-Foster J, Grody WW, Hegde M, Lyon E, Spector E, Voelkerding K, Rehm HL; ACMG Laboratory Quality Assurance Committee. Standards and guidelines for the interpretation of sequence variants: a joint consensus recommendation of the American College of Medical Genetics and Genomics and the Association for Molecular Pathology. Genet Med. 2015 May;17(5):405-24. doi: 10.1038/gim.2015.30. Epub 2015 Mar 5. PMID 25741868
- [Background] MacArthur DG, Manolio TA, Dimmock DP, Rehm HL, Shendure J, Abecasis GR, Adams DR, Altman RB, Antonarakis SE, Ashley EA, Barrett JC, Biesecker LG, Conrad DF, Cooper GM, Cox NJ, Daly MJ, Gerstein MB, Goldstein DB, Hirschhorn JN, Leal SM, Pennacchio LA, Stamatoyannopoulos JA, Sunyaev SR, Valle D, Voight BF, Winckler W, Gunter C. Guidelines for investigating causality of sequence variants in human disease. Nature. 2014 Apr 24;508(7497):469-76. doi: 10.1038/nature13127. PMID 24759409